CLINICAL TRIAL: NCT03871205
Title: A Phase I Study on the Safety and the Efficacy of Personalized Neoantigen-primed Dendritic Cell Vaccines for Refractory Lung Cancer
Brief Title: Neoantigen-primed DC Vaccines Therapy for Refractory Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShenzhenPH BTR-001
Record Dates: First submitted 2019-03-07; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Carcinoma, Non-Small Cell Lung; Carcinoma, Small Cell Lung
Keywords: Neoantigen; Dentritic cell vaccine; Immunotherapy; Refractory lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccinated group (Experimental): Neoantigen loaded-DC vaccination will be performed with 6 doses in total, once per week, adjacent lymph-node injection.
  Interventions: Biological: Neoantigen loaded DC vaccine

INTERVENTIONS:
Biological: Neoantigen loaded DC vaccine — Patients will be vaccinated with autologous mature dendritic cells loaded with neoantigen, DC vaccine will be injected subcutaneously 6 times, once a week.

SUMMARY:
Various of immunotherapies are now widely applied in the treatment of lung cancer. Neoantigens arising from the mutations of the tumor genome expressed specifically on the tumor cell instead of normal cells, suggesting that vaccines targeting neoantigens should generate a highly tumor-specific response with minimal off-target effects. Neoantigens are highly suitable for the development of cancer vaccines. The study aims to evaluate the safety and efficacy of neoantigen-loaded dendritic cell (DC) vaccines for refractory lung cancer.

DETAILED DESCRIPTION:
Cancer genome research has exploded benefits from the application of modern high-throughput genome sequencing in the past few years. Since usually there are no common antigens expressed on the surfaces of different kinds of tumors, neoantigens which expressed specifically in the individual tumor are chosen to establish tumor-specific vaccines.

30 patients with refractory lung cancer would be enrolled and undergo tumor resection if all requirements are met. The whole-exome sequencing and the bioinformatic analysis of the resected specimens would be performed to identify the neoantigens. Then, candidate neoantigens would be synthesized to pulse the matured DC cells. Neoantigen-primed DC vaccines are provided to the corresponding patients. Each patient would be vaccinated 6 times in total, one shot per week.

Patients enrolled would undergo the schemed follow-up, one time per three months. The side effects, overall survival, and progress-free survival would be recorded. At the end of the research, the safety and efficacy of neoantigen DC vaccines for refractory lung cancer would be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years ≤ 70 years at the time of informed consent
* Signed informed consent to be provided
* pathologically confirmed lung cancer
* failed in previous standard chemotherapy and targeted therapy
* Life expectancy not less than 90 days
* Karnofsky performance status 0-1
* adequate organ functions

Exclusion Criteria:

* Actively infectious condition including hepatitis
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Active systemic infections, coagulation disorders or any other active major medical illnesses.
* Patients who are receiving any other investigational agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 3 months after the last vaccination injection
  Safety of personalized neoantigen vaccine will be measured by the number of subjects experiencing each type of adverse event. Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.
Immunogenicity of neoantigen-primed DC Vaccines | once per three month
  Immunogenicity of the DC vaccine will be measured to detect changes of neoantigen-specific T cells by flow cytometry.

SECONDARY OUTCOMES:
Objective Response Rate | once per three months
  The objective response rate is equal to the proportion of participants achieving a best overall response of partial response or complete response (PR + CR). Percentage of Participants Achieving a Stable Disease (SD) or a confirmed CR or PR (Disease Control Rate) Participants achieved disease control if they had a best overall response of CR, PR or SD.
Overall Survival (OS) | through study completion, an average of 1 year
  OS was defined as the time in months from the date of randomization to the date of death from any cause. For participants not known to have died as of the cut-off date, OS was censored at the last known date alive.
Progression-free Survival (PFS) | up to 24 months after last dose of vaccine
  PFS:duration of time from start of treatment to time of progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Lili Ren, Ph.D., Principal Investigator — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No